CLINICAL TRIAL: NCT06529393
Title: The Analgesic Effect of Shoulder Anterior Capsule (SHAC) Block Versus Suprascapular Nerve Block in Arthroscopic Shoulder Surgeries
Brief Title: The Analgesic Effect of (SHAC) Block Versus Suprascapular Nerve Block in Arthroscopic Shoulder Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rana El-sayed Ali Ibrahim, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHAC Block
Record Dates: First submitted 2024-07-15; First posted 2024-07-31 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Shoulder Pain; Postoperative Pain
Keywords: SHAC Block
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: For the SHAC block, with the patient in a beach-chair position and with the arm in extension,With external rotation and abduction,A 21G 10-cm needle will be inserted using an in-plane approach .The tip of the needle will be placed at the space where the nerve has passed .A volume of 15 mL of a mixture of 2% lidocaine (5 mL) and 0.5% levobupivacaine (10 mL) was injected By injecting the pericapsular space, we reach the terminal articular branches indistinctly from their origin.
  For suprascapular nerve block :
  Patients will be placed in lateral position until supraspinatus or infraspinatus muscle contractions were elicited. Following negative aspiration,A 21G 10-cm needle will be inserted using an in-plane approach .The tip of the needle will be placed at the floor of the supraspinatus fossa where the nerve has passed .A volume of 15 mL of a mixture of 2% lidocaine (5 mL) and 0.5% levobupivacaine (10 mL) was injected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHAC block group (Active Comparator): For the SHAC block, with the patient in a beach-chair position and with the arm in extension, the subscapularis muscle is stretched posteriorly and becomes easily visible. With external rotation and abduction, the coracobrachialis and the biceps brachii muscles are displaced, allowing the visualization of the interfascial space between the deep lamina of the deltoid muscle fascia and the superficial lamina of the subscapularis fascia.Once the injection into the fascial space is achieved, the investigators can proceed towards the glenohumeral pericapsular space by crossing the subscapularis muscle with the needle. By injecting the pericapsular space, the investigators reach the terminal articular branches indistinctly from their origin. Furthermore, through the Weitbrecht foramen, a natural capsular foramen between the upper and middle glenohumeral ligaments, we also reach the intra-articular space .
  Interventions: Procedure: SHAC block
- Suprascapular nerve block group (Active Comparator): Patients will be placed in lateral position by using A high - frequency linear ultrasound probe will be placed approximately 2 cm medial to the medial border of the acromion and about 2 cm cranial to the superior margin of the scapular spine until supraspinatus or infraspinatus muscle contractions were elicited. Following negative aspiration,A 21G 10-cm needle will be inserted using an in-plane approach .The tip of the needle will be placed at the floor of the supraspinatus fossa where the nerve has passed .A volume of 15 mL of a mixture of 2% lidocaine (5 mL) and 0.5% levobupivacaine (10 mL) was injected.
  Interventions: Procedure: suprascapular nerve block

INTERVENTIONS:
Procedure: SHAC block — with the patient in a beach-chair position and with the arm in extension, the subscapularis muscle is stretched posteriorly and becomes easily visible. With external rotation and abduction, the coracobrachialis and the biceps brachii muscles are displaced, allowing the visualization of the interfascial space between the deep lamina of the deltoid muscle fascia and the superficial lamina of the subscapularis fascia.Once the injection into the fascial space is achieved, the investigators can proceed towards the glenohumeral pericapsular space by crossing the subscapularis muscle with the needle. By injecting the pericapsular space, the investigators reach the terminal articular branches indistinctly from their origin. Furthermore, through the Weitbrecht foramen, a natural capsular foramen between the upper and middle glenohumeral ligaments, the investigators also reach the intra-articular space .
  Other Names: shoulder anterior capsule block
  Arms: SHAC block group
Procedure: suprascapular nerve block — Patients will be placed in lateral position by using A high - frequency linear ultrasound probe will be placed approximately 2 cm medial to the medial border of the acromion and about 2 cm cranial to the superior margin of the scapular spine until supraspinatus or infraspinatus muscle contractions were elicited. Following negative aspiration,A 21G 10-cm needle will be inserted using an in-plane approach .The tip of the needle will be placed at the floor of the supraspinatus fossa where the nerve has passed .A volume of 15 mL of a mixture of 2% lidocaine (5 mL) and 0.5% levobupivacaine (10 mL) was injected.
  Arms: Suprascapular nerve block group

SUMMARY:
The aim of the study is to compare the post-operative analgesic effect of Shoulder anterior capsule (SHAC) block with Suprascapular nerve block for arthroscopic shoulder surgery with a hypothesis that both Shoulder anterior capsule (SHAC) block and Suprascapular nerve block are effective in providing postoperative analgesia for arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
The role of shoulder arthroscopy in the diagnosis and treatment of shoulder disorders is evolving .

Advances in modern arthroscopy have contributed significantly to greater flexibility and efficacy in addressing shoulder pathology.Advantages of arthroscopy include less invasive approaches, improved visualization, decreased risk of many postoperative complications ,and faster recovery.

Shoulder surgery is well recognised as having the potential to cause severe postoperative pain.The aim of this review is to assess critically the evidence relating to the effectiveness of regional anaesthesia techniques commonly used for postoperative analgesia following shoulder surgery opioid analgesics are commonly used for analgesia when nerve block are not used. opoids are effective in relieving postoperative pain at rest but may increase postoperative nausea and vomiting (PONV),somnolence,constipation,urinary retention,respiratory depression ,and sleep disturbances.

supplementing general anesthesia (GA) with a regional nerve block might improve the quality of postoperative relief pain .

Throughout intraoperative and postoperative period, nerve blocks have been used more populary than others because of efficacy.For the regional nerve block,local anesthetic should be infiltrated close to the nerve for maximum effect.

Shoulder anterior capsule block (SHAC):is combination of two different blocks .the first block is the interfascial space between the deep layer of the deltoid fascia and the superficial layer of the subscapularis fascia , anterior to the subscapularis myotendinous junction . Thanks to this interfascial space,we can reach both the axillary nerve and the subscapular nerves,the lateral pectoral nerve and the musculocutaneous nerve.

Suprascapular nerve block(SSB) :The suprascabular nerve (SSN) originates from the nerve roots and provides sensation for the posterior shoulder capsule, acromioclavicular joint,subacromial bursa,and coracoclavicular ligament .Blocking it provides pre-emptive anesthesia , decreased intraoperative pain ,and postoperative pain relief in shoulder arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* -Age between 18-65 years.
* Body mass index (BMI)of 18-35Kg /m2.
* Patients with American society of anesthesiologist (ASA) physical status | / ||.
* Patients scheduled for elective Arthroscopic Shoulder Surgery.
* Both sexes, males and females.

Exclusion Criteria:

* -Patient refusal.
* Allergy to local anaesthetics.
* Infection at the site of injection .
* Coagulopathy.
* Chronin pain syndromes.
* Prolonged opioid medication

  .-Patients who received any analgesia 24 h before surgery.
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
effect on postopeartive pain after shoulder arthrscopy | baseline
  the pain intensity assessment at rest and on coughing using Numerical Rating Scale (NRS) This will measure pain intensity from 0 to 10 , 0: no pain 3:mild pain 7:moderate pain 10:severe pain

SECONDARY OUTCOMES:
-inceidence of (POVN) 24 hours postoperatively -Block related complications during and after block procedure till 24 hours postoperatively (LAST, pneumohorax and vascular puncture during block procedure) | first 24 hours
  patients complaint from occurrence of nausea and vomiting
-Time of the first opioid request | first 24 hour
  time of the first opioid request , concentration and occurrence of complications (hypotension,bradycardia,itching,urinary retention.) all over 24 hours postoperatively
-Block related complications during and after block procedure till 24 hours postoperatively (LAST, pneumohorax and vascular puncture during block procedure) | first 24 hours
  occurrence of any complications from technical errors

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Hassanen, professor, Study Chair — Assuit university Hospital; Rana EA Ibrahim, Resident, Principal Investigator — Assuit university Hospital; Ayman Abdel Khalek, Ass professor, Study Director — Assuit university Hospital
Locations (1):
- New Trauma Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
method outcome

REFERENCES:
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Background] Paxton ES, Backus J, Keener J, Brophy RH. Shoulder arthroscopy: basic principles of positioning, anesthesia, and portal anatomy. J Am Acad Orthop Surg. 2013 Jun;21(6):332-42. doi: 10.5435/JAAOS-21-06-332. PMID 23728958
- [Background] Singelyn FJ, Lhotel L, Fabre B. Pain relief after arthroscopic shoulder surgery: a comparison of intraarticular analgesia, suprascapular nerve block, and interscalene brachial plexus block. Anesth Analg. 2004 Aug;99(2):589-92, table of contents. doi: 10.1213/01.ANE.0000125112.83117.49. PMID 15271745
- [Background] Basat HC, Ucar DH, Armangil M, Guclu B, Demirtas M. Post operative pain management in shoulder surgery: Suprascapular and axillary nerve block by arthroscope assisted catheter placement. Indian J Orthop. 2016 Nov-Dec;50(6):584-589. doi: 10.4103/0019-5413.193474. PMID 27904211
- [Background] Brenner W, Bohuslavizki KH, Wolf H, Sippel C, Clausen M, Henze E. Radiotherapy with iodine-131 in recurrent malignant struma ovarii. Eur J Nucl Med. 1996 Jan;23(1):91-4. doi: 10.1007/BF01736995. PMID 8586108